CLINICAL TRIAL: NCT01885208
Title: Efficacy and Safety of Semaglutide Once-weekly Versus Exenatide ER 2.0 mg Once-weekly as add-on to 1-2 Oral Antidiabetic Drugs (OADs) in Subjects With Type 2 Diabetes (SUSTAIN™ 3 - vs. QW GLP-1)
Brief Title: Efficacy and Safety of Semaglutide Once-weekly Versus Exenatide ER 2.0 mg Once-weekly as add-on to 1-2 Oral Antidiabetic Drugs (OADs) in Subjects With Type 2 Diabetes
Acronym: SUSTAIN™ 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9535-3624; 2012-004826-92 (EudraCT Number); U1111-1135-8647 (Other: WHO)
Record Dates: First submitted 2013-06-20; First posted 2013-06-24 (Estimated); Results first posted 2018-03-30 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-05

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide; Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Semaglutide 1.0 mg (Experimental)
  Interventions: Drug: semaglutide
- Exenatide ER 2.0 mg (Active Comparator)
  Interventions: Drug: exenatide

INTERVENTIONS:
Drug: semaglutide — One dose of 1.0 mg semaglutide administered subcutaneously (s.c., under the skin) once-weekly
  Arms: Semaglutide 1.0 mg
Drug: exenatide — One dose of 2.0 mg exenatide ER administered subcutaneously (s.c., under the skin) once-weekly
  Other Names: Bydureon®
  Arms: Exenatide ER 2.0 mg

SUMMARY:
This trial is conducted in Europe and North and South America. The aim of the trial is to investigate the efficacy and safety of semaglutide once-weekly versus exenatide ER (extended release) 2.0 mg once-weekly as add-on to 1-2 oral antidiabetic drugs (OADs) in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria: - Subjects diagnosed with type 2 diabetes and on stable diabetes treatment with 1-2 OADs (Metformin equal to or above 1500 mg or maximum tolerated dose and/or thiazolidinedione (TZD) and sulfonylureas (SUs) equal to or above half of maximum dose allowed according to national label) for at least 90 days prior to screening. Stable is defined as unchanged medication and unchanged dose - HbA1c 7.0 - 10.5 % (53 - 91 mmol/mol) (both inclusive) Exclusion Criteria: - Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using an adequate contraceptive method throughout the trial including the 5 week follow-up period (adequate contraceptive measures as required by local law or practice) - Any chronic disorder or severe disease which, in the opinion of the investigator, might jeopardise subject's safety or compliance with the protocol - Treatment with glucose lowering agent(s) other than stated in the inclusion criteria in a period of 90 days before screening. An exception is short-term treatment (7 days or less in total) with insulin in connection with inter-current illness - History of chronic or idiopathic acute pancreatitis - Screening calcitonin value equal to or above 50 ng/L (pg/mL) - Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN 2) - Impaired renal function defined as estimated glomerular filtration rate (eGFR) below 60 ml/min/1.73 m^2 per modification of diet in renal disease (MDRD) formula (4 variable version) - Acute coronary or cerebrovascular event within 90 days before randomisation - Heart failure, New York Heart Association (NYHA) class IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 813 (Actual)
Dates: Start 2013-12-02 (Actual); Primary Completion 2015-07-13 (Actual); Study Completion 2015-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (126):
- United States (64):
  - Novo Nordisk Investigational Site, Anniston, Alabama
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Pell City, Alabama
  - Novo Nordisk Investigational Site, Glendale, Arizona
  - Novo Nordisk Investigational Site, Mesa, Arizona
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Burbank, California
  - Novo Nordisk Investigational Site, Hawaiian Gardens, California
  - Novo Nordisk Investigational Site, Lomita, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Northridge, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, Tustin, California
  - Novo Nordisk Investigational Site, Colorado Springs, Colorado
  - Novo Nordisk Investigational Site, Bradenton, Florida
  - Novo Nordisk Investigational Site, Brandon, Florida
  - Novo Nordisk Investigational Site, Coral Gables, Florida
  - Novo Nordisk Investigational Site, Hialeah, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Miami Lakes, Florida
  - Novo Nordisk Investigational Site, Plantation, Florida
  - Novo Nordisk Investigational Site, Savannah, Georgia
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Franklin, Indiana
  - Novo Nordisk Investigational Site, Greenfield, Indiana
  - Novo Nordisk Investigational Site, Muncie, Indiana
  - Novo Nordisk Investigational Site, Louisville, Kentucky
  - Novo Nordisk Investigational Site, Madisonville, Kentucky
  - Novo Nordisk Investigational Site, Hyattsville, Maryland
  - Novo Nordisk Investigational Site, Kalamazoo, Michigan
  - Novo Nordisk Investigational Site, St Louis, Missouri
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Mine Hill, New Jersey
  - Novo Nordisk Investigational Site, Albuquerque, New Mexico
  - Novo Nordisk Investigational Site, North Massapequa, New York
  - Novo Nordisk Investigational Site, Syracuse, New York
  - Novo Nordisk Investigational Site, West Seneca, New York
  - Novo Nordisk Investigational Site, Greensboro, North Carolina
  - Novo Nordisk Investigational Site, Hickory, North Carolina
  - Novo Nordisk Investigational Site, Whiteville, North Carolina
  - Novo Nordisk Investigational Site, Akron, Ohio
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Cleveland, Ohio
  - Novo Nordisk Investigational Site, Delaware, Ohio
  - Novo Nordisk Investigational Site, Corvallis, Oregon
  - Novo Nordisk Investigational Site, Portland, Oregon
  - Novo Nordisk Investigational Site, Lansdale, Pennsylvania
  - Novo Nordisk Investigational Site, Norristown, Pennsylvania
  - Novo Nordisk Investigational Site, Charleston, South Carolina
  - Novo Nordisk Investigational Site, Mt. Pleasant, South Carolina
  - Novo Nordisk Investigational Site, Murrells Inlet, South Carolina
  - Novo Nordisk Investigational Site, Spartanburg, South Carolina
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Austin, Texas
  - Novo Nordisk Investigational Site, Carrollton, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Fort Worth, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Irving, Texas
  - Novo Nordisk Investigational Site, Katy, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Sugar Land, Texas
  - Novo Nordisk Investigational Site, Alexandria, Virginia
- Argentina (4):
  - Novo Nordisk Investigational Site, Buenos Aires
  - Novo Nordisk Investigational Site, CABA
  - Novo Nordisk Investigational Site, Lanús Este
  - Novo Nordisk Investigational Site, Mar del Plata
- Croatia (5):
  - Novo Nordisk Investigational Site, Karlovac
  - Novo Nordisk Investigational Site, Osijek
  - Novo Nordisk Investigational Site, Slavonski Brod
  - Novo Nordisk Investigational Site, Virovitica
  - Novo Nordisk Investigational Site, Zagreb
- Finland (4):
  - Novo Nordisk Investigational Site, Helsinki
  - Novo Nordisk Investigational Site, Kerava
  - Novo Nordisk Investigational Site, Oulu
  - Novo Nordisk Investigational Site, Turku
- France (8):
  - Novo Nordisk Investigational Site, Châlons-en-Champagne
  - Novo Nordisk Investigational Site, Corbeil-Essonnes
  - Novo Nordisk Investigational Site, La Rochelle
  - Novo Nordisk Investigational Site, Le Creusot
  - Novo Nordisk Investigational Site, Nanterre
  - Novo Nordisk Investigational Site, Roubaix
  - Novo Nordisk Investigational Site, Strasbourg
  - Novo Nordisk Investigational Site, Vénissieux
- Germany (7):
  - Novo Nordisk Investigational Site, Dresden
  - Novo Nordisk Investigational Site, Duisburg
  - Novo Nordisk Investigational Site, Hohenmölsen
  - Novo Nordisk Investigational Site, Mannheim
  - Novo Nordisk Investigational Site, Oldenburg
  - Novo Nordisk Investigational Site, Rehlingen-Siersburg
  - Novo Nordisk Investigational Site, Völklingen
- Greece (3):
  - Novo Nordisk Investigational Site, Athens
  - Novo Nordisk Investigational Site, Piraeus
  - Novo Nordisk Investigational Site, Thessaloniki
- Italy (7):
  - Novo Nordisk Investigational Site, Bologna
  - Novo Nordisk Investigational Site, Città di Castello
  - Novo Nordisk Investigational Site, Milan
  - Novo Nordisk Investigational Site, Palermo
  - Novo Nordisk Investigational Site, Pavia
  - Novo Nordisk Investigational Site, Roma
  - Novo Nordisk Investigational Site, Siena
- Netherlands (8):
  - Novo Nordisk Investigational Site, Amsterdam
  - Novo Nordisk Investigational Site, Apeldoorn
  - Novo Nordisk Investigational Site, Delft
  - Novo Nordisk Investigational Site, Hoofddorp
  - Novo Nordisk Investigational Site, Leeuwarden
  - Novo Nordisk Investigational Site, Rotterdam
  - Novo Nordisk Investigational Site, Venlo
  - Novo Nordisk Investigational Site, Zoetermeer
- Puerto Rico (2):
  - Novo Nordisk Investigational Site, Caguas
  - Novo Nordisk Investigational Site, Manatí
- Serbia (3):
  - Novo Nordisk Investigational Site, Belgrade
  - Novo Nordisk Investigational Site, Kragujevac
  - Novo Nordisk Investigational Site, Novi Sad
- Switzerland (5):
  - Novo Nordisk Investigational Site, Basel
  - Novo Nordisk Investigational Site, Geneva
  - Novo Nordisk Investigational Site, Lucerne
  - Novo Nordisk Investigational Site, Sankt Gallen
  - Novo Nordisk Investigational Site, Zollikerberg
- United Kingdom (6):
  - Novo Nordisk Investigational Site, Ayr
  - Novo Nordisk Investigational Site, Bath
  - Novo Nordisk Investigational Site, Bradford-on-Avon
  - Novo Nordisk Investigational Site, Haxey
  - Novo Nordisk Investigational Site, Headington
  - Novo Nordisk Investigational Site, Rotherham

REFERENCES:
- [Background] Fonseca VA, Capehorn MS, Garg SK, Jodar Gimeno E, Hansen OH, Holst AG, Nayak G, Seufert J. Reductions in Insulin Resistance are Mediated Primarily via Weight Loss in Subjects With Type 2 Diabetes on Semaglutide. J Clin Endocrinol Metab. 2019 Sep 1;104(9):4078-4086. doi: 10.1210/jc.2018-02685. PMID 30938762
- [Background] Rodbard HW, Bellary S, Hramiak I, Seino Y, Silver R, Damgaard LH, Nayak G, Zacho J, Aroda VR. GREATER COMBINED REDUCTIONS IN HbA1C >/=1.0% AND WEIGHT >/=5.0% WITH SEMAGLUTIDE VERSUS COMPARATORS IN TYPE 2 DIABETES. Endocr Pract. 2019 Jun;25(6):589-597. doi: 10.4158/EP-2018-0444. Epub 2019 Mar 13. PMID 30865526
- [Result] Ahmann AJ, Capehorn M, Charpentier G, Dotta F, Henkel E, Lingvay I, Holst AG, Annett MP, Aroda VR. Efficacy and Safety of Once-Weekly Semaglutide Versus Exenatide ER in Subjects With Type 2 Diabetes (SUSTAIN 3): A 56-Week, Open-Label, Randomized Clinical Trial. Diabetes Care. 2018 Feb;41(2):258-266. doi: 10.2337/dc17-0417. Epub 2017 Dec 15. PMID 29246950
- [Result] Warren M, Chaykin L, Trachtenbarg D, Nayak G, Wijayasinghe N, Cariou B. Semaglutide as a therapeutic option for elderly patients with type 2 diabetes: Pooled analysis of the SUSTAIN 1-5 trials. Diabetes Obes Metab. 2018 Sep;20(9):2291-2297. doi: 10.1111/dom.13331. Epub 2018 Jun 7. PMID 29687620
- [Result] Petri KCC, Ingwersen SH, Flint A, Zacho J, Overgaard RV. Exposure-response analysis for evaluation of semaglutide dose levels in type 2 diabetes. Diabetes Obes Metab. 2018 Sep;20(9):2238-2245. doi: 10.1111/dom.13358. Epub 2018 Jun 15. PMID 29748996
- [Result] Ahren B, Atkin SL, Charpentier G, Warren ML, Wilding JPH, Birch S, Holst AG, Leiter LA. Semaglutide induces weight loss in subjects with type 2 diabetes regardless of baseline BMI or gastrointestinal adverse events in the SUSTAIN 1 to 5 trials. Diabetes Obes Metab. 2018 Sep;20(9):2210-2219. doi: 10.1111/dom.13353. Epub 2018 Jun 12. PMID 29766634
- [Result] DeVries JH, Desouza C, Bellary S, Unger J, Hansen OKH, Zacho J, Woo V. Achieving glycaemic control without weight gain, hypoglycaemia, or gastrointestinal adverse events in type 2 diabetes in the SUSTAIN clinical trial programme. Diabetes Obes Metab. 2018 Oct;20(10):2426-2434. doi: 10.1111/dom.13396. Epub 2018 Jul 9. PMID 29862621
- [Result] Carlsson Petri KC, Ingwersen SH, Flint A, Zacho J, Overgaard RV. Semaglutide s.c. Once-Weekly in Type 2 Diabetes: A Population Pharmacokinetic Analysis. Diabetes Ther. 2018 Aug;9(4):1533-1547. doi: 10.1007/s13300-018-0458-5. Epub 2018 Jun 15. PMID 29907893
- [Result] Malkin SJP, Russel-Szymczyk M, Liidemann G, Volke V, Hunt B. Once-Weekly Semaglutide Versus Once-Daily Liraglutide for the Treatment of Type 2 Diabetes: A Long-Term Cost-Effectiveness Analysis in Estonia. Diabetes Ther. 2019 Feb;10(1):159-176. doi: 10.1007/s13300-018-0542-x. Epub 2018 Dec 7. PMID 30535837
- [Result] Aroda VR, Ahmann A, Cariou B, Chow F, Davies MJ, Jodar E, Mehta R, Woo V, Lingvay I. Comparative efficacy, safety, and cardiovascular outcomes with once-weekly subcutaneous semaglutide in the treatment of type 2 diabetes: Insights from the SUSTAIN 1-7 trials. Diabetes Metab. 2019 Oct;45(5):409-418. doi: 10.1016/j.diabet.2018.12.001. Epub 2019 Jan 4. PMID 30615985
- [Result] Overgaard RV, Lindberg SO, Thielke D. Impact on HbA1c and body weight of switching from other GLP-1 receptor agonists to semaglutide: A model-based approach. Diabetes Obes Metab. 2019 Jan;21(1):43-51. doi: 10.1111/dom.13479. Epub 2018 Aug 23. PMID 30047216
- [Derived] Mosenzon O, Capehorn MS, De Remigis A, Rasmussen S, Weimers P, Rosenstock J. Impact of semaglutide on high-sensitivity C-reactive protein: exploratory patient-level analyses of SUSTAIN and PIONEER randomized clinical trials. Cardiovasc Diabetol. 2022 Sep 2;21(1):172. doi: 10.1186/s12933-022-01585-7. PMID 36056351
- [Derived] Husain M, Bain SC, Holst AG, Mark T, Rasmussen S, Lingvay I. Effects of semaglutide on risk of cardiovascular events across a continuum of cardiovascular risk: combined post hoc analysis of the SUSTAIN and PIONEER trials. Cardiovasc Diabetol. 2020 Sep 30;19(1):156. doi: 10.1186/s12933-020-01106-4. PMID 32998732
- [Derived] Lingvay I, Capehorn MS, Catarig AM, Johansen P, Lawson J, Sandberg A, Shaw R, Paine A. Efficacy of Once-Weekly Semaglutide vs Empagliflozin Added to Metformin in Type 2 Diabetes: Patient-Level Meta-analysis. J Clin Endocrinol Metab. 2020 Dec 1;105(12):e4593-604. doi: 10.1210/clinem/dgaa577. PMID 32827435
- [Derived] Capehorn M, Ghani Y, Hindsberger C, Johansen P, Jodar E. Once-Weekly Semaglutide Reduces HbA1c and Body Weight in Patients with Type 2 Diabetes Regardless of Background Common OAD: a Subgroup Analysis from SUSTAIN 2-4 and 10. Diabetes Ther. 2020 May;11(5):1061-1075. doi: 10.1007/s13300-020-00796-z. Epub 2020 Mar 19. PMID 32193837
- [Derived] Husain M, Bain SC, Jeppesen OK, Lingvay I, Sorrig R, Treppendahl MB, Vilsboll T. Semaglutide (SUSTAIN and PIONEER) reduces cardiovascular events in type 2 diabetes across varying cardiovascular risk. Diabetes Obes Metab. 2020 Mar;22(3):442-451. doi: 10.1111/dom.13955. Epub 2020 Feb 5. PMID 31903692
- [Derived] DeSouza C, Cariou B, Garg S, Lausvig N, Navarria A, Fonseca V. Efficacy and Safety of Semaglutide for Type 2 Diabetes by Race and Ethnicity: A Post Hoc Analysis of the SUSTAIN Trials. J Clin Endocrinol Metab. 2020 Feb 1;105(2):dgz072. doi: 10.1210/clinem/dgz072. PMID 31769496
- [Derived] Jendle J, Birkenfeld AL, Polonsky WH, Silver R, Uusinarkaus K, Hansen T, Hakan-Bloch J, Tadayon S, Davies MJ. Improved treatment satisfaction in patients with type 2 diabetes treated with once-weekly semaglutide in the SUSTAIN trials. Diabetes Obes Metab. 2019 Oct;21(10):2315-2326. doi: 10.1111/dom.13816. Epub 2019 Jul 12. PMID 31215727
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of 146 sites selected for recruitment, 138 sites in 12 countries randomised subjects to the treatment viz. Argentina: 4 sites; Croatia: 5 sites; Finland: 5 sites; France: 7 sites; Germany: 7 sites; Greece: 5 sites; Italy: 6 sites; Netherlands: 8 sites; Serbia: 5 sites; Switzerland: 5 sites; United Kingdom: 6 sites and United States: 75 sites
Groups:
- Semaglutide 1.0 mg: Subjects randomised to semaglutide followed a fixed dose-escalation regimen for a period of 56 weeks. Subjects started with once-weekly doses of 0.25 mg for 4 weeks, then escalated to doses of 0.5 mg once weekly for 4 weeks, and finally escalated to 1.0 mg once weekly (maximum dose). Doses were not changed during the trial after the maintenance dose was reached. Semaglutide 1.34 mg/mL was supplied in a 1.5 mL pre-filled PDS290 pen-injector and was to be administered subcutaneously (s.c.; under the skin) either in the thigh, abdomen or upper arm at the same weekday. All subjects continued their pre-trial treatment of 1-2 oral anti-diabetes drug (OAD) therapy throughout the trial, unless rescue medication was needed.
- Exenatide ER 2.0 mg: Subjects on exenatide extended release (ER) 2.0 mg (Bydureon®) were treated with the same 2.0 mg dose for a period of 56 weeks. Exenatide one vial of 2 mg exenatide ER was supplied in a pre-filled syringe of 0.65 mL solvent and to be administrated subcutaneously (s.c.; under the skin) once weekly through out the trial. All subjects continued their pre-trial treatment of 1-2 OAD therapy entire trial, unless rescue medication was needed.
Period: Overall Study
Arm/Group | Semaglutide 1.0 mg | Exenatide ER 2.0 mg
Started | 406 | 407
Exposed | 404 | 405
Premature Discontinuation of Treatment | 82 (Subjects who prematurely discontinued treatment were allowed to continue participation in the trial.) | 85 (Subjects who prematurely discontinued treatment were allowed to continue participation in the trial.)
Completed | 374 | 369
Not Completed | 32 | 38
Not completed — Unclassified | 32 | 38

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomised subjects who have received at least one dose of randomised semaglutide 1.0 mg or exenatide ER 2.0 mg. Subjects in the FAS contributed to the evaluation based on the treatment assigned at randomisation.
Groups:
- Exenatide ER 2.0 mg: Subjects randomised to exenatide extended release (ER) 2.0 mg (Bydureon®) were treated with the same 2.0 mg dose for a period of 56 weeks. Exenatide one vial of 2 mg exenatide ER was supplied in a pre-filled syringe of 0.65 mL solvent and to be administrated subcutaneously (s.c.; under the skin) once weekly through out the trial. All subjects continued their pre-trial treatment of 1-2 OAD therapy entire trial, unless rescue medication was needed.
- Total: Total of all reporting groups
Arm/Group | Semaglutide 1.0 mg | Exenatide ER 2.0 mg | Total
Number analyzed (Participants) | 404 | 405 | 809
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (10.3) | 56.7 (11.1) | 56.6 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 185 | 177 | 362
  Male | 219 | 228 | 447
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.36 (0.95) | 8.33 (0.96) | 8.35 (0.95)
Body Weight [Mean (Standard Deviation); unit: kilogram (s)] | 96.21 (22.5) | 95.37 (20.46) | 95.79 (21.49)
Fasting Plasma Glucose [Mean (Standard Deviation); unit: mg/ dL] — Population: The number of subjects analysed in the semaglutide and exenatide arms was 383 and 384, respectively.
  mg/ dL
    number analyzed (Participants) | 383 | 384 | 767
    (all) | 190.5 (48.06) | 187.5 (49.41) | 189.0 (48.74)
Systolic blood pressure [Mean (Standard Deviation); unit: mm Hg] — Population: The number of subjects analysed in the semaglutide and exenatide arms was 404 and 404, respectively.
  mm Hg
    number analyzed (Participants) | 404 | 404 | 808
    (all) | 133.35 (14.87) | 133.66 (14.25) | 133.51 (14.55)
Diastolic blood pressure [Mean (Standard Deviation); unit: mm Hg] — Population: The number of subjects analysed in the semaglutide and exenatide arms was 404 and 404, respectively.
  mm Hg
    number analyzed (Participants) | 404 | 404 | 808
    (all) | 80.23 (8.67) | 79.57 (8.8) | 79.90 (8.73)
Patient-reported outcome: Diabetes Treatment Satisfaction Questionnaire (DTSQ) [Mean (Standard Deviation); unit: Units on a scale] — The DTSQs was used to assess a subject's treatment satisfaction. This questionnaire contained 8 components and measures the treatment for diabetes (including insulin, tablets and/or diet) in terms of convenience, flexibility and general feelings regarding treatment. The value presented is the 'Treatment Satisfaction' summary score, which is the sum of 6 of the 8 items of the DTSQs questionnaire. Response options range from 6 (best case) to 0 (worst case). Total scores for treatment satisfaction range from 0-36. Higher scores indicate higher satisfaction. Population: The number of subjects analysed in the semaglutide and exenatide arms was 403 and 405, respectively.
  Units on a scale
    number analyzed (Participants) | 403 | 405 | 808
    (all) | 27.35 (6.55) | 27.23 (6.62) | 27.29 (6.58)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c (Glycosylated Haemoglobin)
Description: Mean change in HbA1c from baseline to week 56.
Time Frame: Week 0, week 56
Population: The full analysis set (FAS) included all randomised subjects who had received at least one dose of randomised semaglutide 1.0 mg or exenatide ER 2.0 mg.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated haemoglobin
Arm/Group | Semaglutide 1.0 mg | Exenatide ER 2.0 mg
Number analyzed (Participants) | 404 | 405
percentage of glycosylated haemoglobin | -1.54 (0.06) | -0.92 (0.06)
Statistical Analysis 1: Comparison: Semaglutide 1.0 mg vs Exenatide ER 2.0 mg; The post-baseline responses were analysed using a mixed model for repeated measurements with treatment and country as fixed factors and baseline value as covariate, all nested within visit; Test type: Non-Inferiority — Non-inferiority was concluded if the upper limit of the two-sided 95% confidence interval for the estimated treatment difference between semaglutide 1.0 mg and exenatide ER 2.0 mg was below the pre-specified non-inferiority margin (0.3 %); p < 0.0001, Mixed Models Analysis; Treatment difference = -0.62, 95% CI 2-sided [-0.8 to -0.44]
Statistical Analysis 2: Comparison: Semaglutide 1.0 mg vs Exenatide ER 2.0 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — Superiority was concluded if the upper limit of the two-sided 95% confidence interval for the estimated treatment difference between semaglutide 1.0 mg and exenatide ER 2.0 mg was below the pre-specified superiority margin (0 %); p < 0.0001, Mixed Models Analysis; Treatment difference = -0.62, 95% CI 2-sided [-0.8 to -0.44]

2. Secondary Outcome: Change From Baseline in Body Weight
Description: Mean change in body weight from baseline to week 56.
Time Frame: Week 0, week 56
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kilograms
Arm/Group | Semaglutide 1.0 mg | Exenatide ER 2.0 mg
Number analyzed (Participants) | 404 | 405
kilograms | -5.63 (0.29) | -1.85 (0.29)

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG)
Description: Mean change in FPG from baseline to week 56.
Time Frame: Week 0, week 56
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Semaglutide 1.0 mg | Exenatide ER 2.0 mg
Number analyzed (Participants) | 404 | 405
mg/dL | -51.22 (2.36) | -36.1 (2.45)

4. Secondary Outcome: Change From Baseline in Systolic and Diastolic Blood Pressure
Description: Mean changes in systolic and diastolic blood pressure from baseline to week 56.
Time Frame: Week 0, week 56
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Semaglutide 1.0 mg | Exenatide ER 2.0 mg
Number analyzed (Participants) | 404 | 405
mm Hg
  Systolic blood pressure: number analyzed (Participants) | 295 | 275
  Systolic blood pressure | -4.6 (0.68) | -2.23 (0.7)
  Diastolic blood pressure: number analyzed (Participants) | 295 | 275
  Diastolic blood pressure | -1.0 (0.45) | -0.1 (0.46)

5. Secondary Outcome: Change From Baseline in Patient Reported Outcome (PRO) Questionnaire Diabetes Treatment Satisfaction Questionnaire Status (DTSQs)
Description: The Diabetes Treatment Satisfaction Questionnaire (DTSQs) was used to assess a subject's treatment satisfaction. This questionnaire contained 8 components and measures the treatment for diabetes (including insulin, tablets and/or diet) in terms of convenience, flexibility and general feelings regarding treatment. The value presented is the 'Treatment Satisfaction' summary score, which is the sum of 6 of the 8 items of the DTSQs questionnaire. Response options range from 6 (best case) to 0 (worst case). Total scores for treatment satisfaction range from 0-36. Higher scores indicate higher satisfaction.
Time Frame: Week 0, week 56
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Semaglutide 1.0 mg | Exenatide ER 2.0 mg
Number analyzed (Participants) | 404 | 405
Units on a scale | 4.98 (0.26) | 3.96 (0.27)

6. Secondary Outcome: Subjects Who Achieve HbA1c Equal to or Below 6.5% (48 mmol/Mol) American Association of Clinical Endocrinologists (AACE) Target: (Yes/no)
Description: The endpoint considered HbA1c ≤6.5% (48 mmol/mol) as per the AACE target after 56 weeks of treatment.
Time Frame: After 56 weeks' treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 1.0 mg | Exenatide ER 2.0 mg
Number analyzed (Participants) | 404 | 405
Participants
  Yes | 190 | 89
  No | 214 | 316

ADVERSE EVENTS:
Time Frame: All adverse events are treatment-emergent adverse events (TEAEs). A TEAE included events that had onset date (or increase in severity) on or after the first day of exposure (week 0) to randomised treatment (week 0-56 treatment period) and no later than the date of last dose + 42 days of follow-up.
Description: The safety analysis set (SAS) included all randomised subjects who have received at least one dose of randomised semaglutide 1.0 mg or exenatide ER 2.0 mg. Subjects in the SAS contributed to the evaluation based on the treatment actually received.
Groups:
- Sema 1.0 mg: Subjects randomised to semaglutide followed a fixed dose-escalation regimen for a period of 56 weeks. Subjects started with once-weekly doses of 0.25 mg for 4 weeks, then escalated to doses of 0.5 mg once weekly for 4 weeks, and finally escalated to 1.0 mg once weekly (maximum dose). Doses were not changed during the trial after the maintenance dose was reached. Semaglutide 1.34 mg/mL was supplied in a 1.5 mL pre-filled PDS290 pen-injector and was to be administered subcutaneously (s.c.; under the skin) either in the thigh, abdomen or upper arm at the same weekday. All subjects continued their pre-trial treatment of 1-2 oral anti-diabetes drug (OAD)therapy throughout the trial, unless rescue medication was needed.
- Exenatide ER: Subjects randomised to exenatide extended release (ER) 2.0 mg(Bydureon®) were treated with the same 2.0 mg dose for a period of 56 weeks. Exenatide one vial of 2 mg exenatide ER was supplied in a pre-filled syringe of 0.65 mL solvent and to be administrated subcutaneously (s.c.; under the skin) once weekly through out the trial. All subjects continued their pre-trial treatment of 1-2 OAD therapy entire trial, unless rescue medication was needed.
Arm/Group | Sema 1.0 mg | Exenatide ER
Serious Adverse Events (participants affected / at risk) | 38/404 | 24/405
Other Adverse Events (participants affected / at risk) | 194/404 | 187/405
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sema 1.0 mg (N=404) | Exenatide ER (N=405)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abortion induced (Surgical and medical procedures) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 3 (3)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Cardiac ablation (Surgical and medical procedures) | 1 (1) | 0 (0)
Castleman's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Coronary arterial stent insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Coronary artery bypass (Surgical and medical procedures) | 2 (2) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2)
Glycosuria (Renal and urinary disorders) | 1 (1) | 0 (0)
HIV test positive (Investigations) | 1 (1) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0)
Meniscus removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Surgical failure (General disorders) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sema 1.0 mg (N=404) | Exenatide ER (N=405)
Constipation (Gastrointestinal disorders) | 26 (28) | 21 (26)
Decreased appetite (Metabolism and nutrition disorders) | 32 (34) | 21 (24)
Diarrhoea (Gastrointestinal disorders) | 46 (86) | 34 (58)
Dyspepsia (Gastrointestinal disorders) | 27 (33) | 19 (23)
Headache (Nervous system disorders) | 38 (81) | 39 (65)
Injection site nodule (General disorders) | 0 (0) | 49 (55)
Lipase increased (Investigations) | 41 (51) | 49 (64)
Nasopharyngitis (Infections and infestations) | 39 (46) | 38 (51)
Nausea (Gastrointestinal disorders) | 90 (159) | 48 (70)
Vomiting (Gastrointestinal disorders) | 29 (37) | 25 (40)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
"At the end of the trial, one or more scientific publications may be prepared collaboratively by the Investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for less than 60 days to protect intellectual property".